CLINICAL TRIAL: NCT00002790
Title: A PHASE I/II STUDY OF RAPAMYCIN (SIROLIMUS) IN COMBINATION WITH METHOTREXATE (MTX) AND CYCLOSPORINE (CPS) IN PATIENTS UNDERGOING MARROW TRANSPLANTATION FROM RELATED DONORS MISMATCHED FOR ONE HLA ANTIGEN IN THE DIRECTION OF GRAFT-VERSUS-HOST DISEASE (GVHD)
Brief Title: Prevention of Graft-Versus-Host Disease in Patients With Hematologic Malignancies Who Are Receiving a Bone Marrow Transplant
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Supportive Care
Other Study IDs: 1096.00; FHCRC-1096.00; NCI-H96-0928; CDR0000064855 (Registry Identifier: PDQ)
Record Dates: First submitted 1999-11-01; First posted 2004-09-02 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Graft Versus Host Disease; Leukemia; Myelodysplastic Syndromes
Keywords: childhood acute lymphoblastic leukemia; chronic lymphocytic leukemia; adult acute lymphoblastic leukemia; adult acute myeloid leukemia; chronic myelogenous leukemia; childhood acute myeloid leukemia/other myeloid malignancies; myelodysplastic syndromes; graft versus host disease; childhood myelodysplastic syndromes
MeSH Terms: conditions — Graft vs Host Disease; Leukemia; Myelodysplastic Syndromes; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myeloid, Acute; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Cyclosporine; Methotrexate; Sirolimus

INTERVENTIONS:
Drug: cyclosporine
Drug: methotrexate
Drug: sirolimus

SUMMARY:
RATIONALE: Bone marrow transplantation may be able to replace immune cells that were destroyed by chemotherapy used to kill tumor cells. Sometimes the transplanted cells can make an immune response against the body's normal tissues. Treatment with sirolimus, methotrexate, and cyclosporine may prevent this from happening.

PURPOSE: Phase I/II trial to study the effectiveness of sirolimus plus methotrexate and cyclosporine in preventing graft-versus-host disease in patients with hematologic malignancies who are receiving a bone marrow transplant.

DETAILED DESCRIPTION:
OBJECTIVES: I. Estimate the maximum tolerated dose of rapamycin that can be safely combined with standard methotrexate/cyclosporine prophylaxis for graft-versus-host disease (GVHD) in patients with hematologic disorders who have received a bone marrow transplant from a related donor who is mismatched for 1 HLA-A, -B, or -DR antigen in the GVHD direction.

OUTLINE: This is a dose escalation study. Groups of 6-12 patients receive escalating doses of rapamycin until the maximum tolerated dose of rapamycin given in combination with methotrexate/cyclosporine is determined. All patients receive cyclosporine from the day prior to transplant until day 50 post-transplant; the dose is then tapered over 130 days. Methotrexate is given on days 1, 3, and 6 post-transplant. Rapamycin is given every other day, days 7-59. Bone marrow transplantation occurs on day 0. Patients may not receive concurrent therapy with agents that could interfere with rapamycin metabolism, intravenous lipids, FK506 or other immunosuppressive agents (prednisone allowed), NSAIDs, or other cytotoxic agents. Patients are followed at 6 months for 2 years, then annually.

PROJECTED ACCRUAL: 12-36 patients will be accrued over 1-2.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: See General Eligibility Criteria

PATIENT CHARACTERISTICS: Age: 13 and over Performance status: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Creatinine no greater than 2.0 mg/dL Cardiovascular: No cardiac disease No clinically significant cardiac abnormality No ischemia No recent injury on EKG Other: No intolerance or unresponsiveness to rapamycin No hypersensitivity to macrolide antibiotics, e.g., erythromycin, azithromycin, clarithromycin No requirement for medications that may significantly affect rapamycin metabolism, i.e.: Carbamazepine Ketoconazole Primidone Cimetidine Nicardipine Rifampin Diltiazem Phenobarbital Valproic acid Erythromycin Phenytoin Verapamil No uncontrolled systemic infection No pregnant or nursing women Negative pregnancy test required of fertile women Effective contraception required of fertile patients during and for 3 months after study Able to tolerate less than 400 mL of liquid oral intake

PRIOR CONCURRENT THERAPY: At least 1 week since any investigational drug

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 1996-03

CONTACTS AND LOCATIONS:
Overall Officials: H. Joachim Deeg, MD, Study Chair — Fred Hutchinson Cancer Center